CLINICAL TRIAL: NCT06796413
Title: Loop Resection or Cold-cup Biopsy? A Prospective Randomized Study Evaluating the Accuracy of Detrusor Muscle Representation During Transurethral Resection of Bladder Tumors
Brief Title: Loop Resection or Cold-cup Biopsy? A Study Comparing the Accuracy of Muscle Samples During Bladder Tumor Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Stellenbosch (Other)
Responsible Party: Principal Investigator, Dr Eduan Delport, Urology Resident, University of Stellenbosch
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 17234
Record Dates: First submitted 2025-01-15; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Bladder Cancer; Bladder Cancer Stage I; TURBT
Keywords: Bladder Cancer; Detrusor Muscle Sampling; Detrusor Muscle Representation; Loop Resection; Cold-Cup Biopsy; Artifacts
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cold-Cup Biopsy (Active Comparator): Cold-Cup Biopsy of bladder tumor base
  Interventions: Procedure: Loop Resection or Cold-cup biopsy
- Loop Resection of bladder tumor base (Experimental): Loop Resection of bladder tumor base
  Interventions: Procedure: Loop Resection or Cold-cup biopsy

INTERVENTIONS:
Procedure: Loop Resection or Cold-cup biopsy — Loop Resection or cold-cup biopsy of bladder tumor base - thus after the tumor has been resected and the deep muscle specimen needed to be obtained, the Loop Cautery or Lowsley Forceps (for cold-cup biopsy) was used to obtain the deep muscle specimen
  Other Names: Loop Cautery; Cold-cup Biopsy

SUMMARY:
In this report the investigators compared two deep muscle sampling methods (Loop resection and Cold-Cup Biopsy) during endoscopic resection of bladder tumors for patients with suspected bladder cancer in Tygerberg hospital. The investigators found that both sampling methods are equal effective with regards to muscle representation, regardless of surgeon experience. An important finding is that Loop Resection produced less tissue artefacts in the deep muscle specimen for the more experienced surgeons, while there was no difference for less experienced surgeons. The investigators thus conclude that - from a practical point of view - Loop Resection should be the deep muscle sampling method of choice.

ELIGIBILITY:
Inclusion Criteria:

* • All patients requiring cystoscopy plus loop resection of bladder tumor.

Exclusion Criteria:

* • Patients who underwent cystoscopy and no loop resection

  * Patients who underwent cystoscopy and only cold-cup biopsy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-07-14 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Detrusor Muscle Representation | From enrollment to the end of treatment at 2-4 weeks when histology results are available
  Histopathological confirmation of detrusor muscle representation in the Deep Muscle Specimen obtained by either the Loop Resection method or Cold-Cup Biopsy method

CONTACTS AND LOCATIONS:
Overall Officials: Eduan Delport, MB, ChB, Principal Investigator — University of Stellenbosch
Locations (1):
- Stellenbosch University - Faculty of Health Sciences - Department of Urology, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: Undecided
Some of the personal detail of the participants may have changed or may not be so easily attainable.